CLINICAL TRIAL: NCT04484623
Title: A Phase III, Multicenter, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of Belantamab Mafodotin in Combination With Pomalidomide and Dexamethasone (B-Pd) Versus Pomalidomide Plus Bortezomib and Dexamethasone (PVd) in Participants With Relapsed/Refractory Multiple Myeloma (DREAMM 8)
Brief Title: Belantamab Mafodotin Plus Pomalidomide and Dexamethasone (Pd) Versus Bortezomib Plus Pd in Relapsed/Refractory Multiple Myeloma
Acronym: DREAMM 8
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 207499; 2018-004354-21 (EudraCT Number)
Expanded Access: NCT03763370 (Available)
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Global Cohort; Belantamab Mafodotin; Relapsed/Refractory Multiple Myeloma; Pomalidomide; Dexamethasone; Bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — belantamab mafodotin; pomalidomide; Dexamethasone; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Belantamab mafodotin plus Pomalidomide and Dexamethasone (Experimental)
  Interventions: Drug: Belantamab mafodotin; Drug: Pomalidomide; Drug: Dexamethasone
- Arm B: Bortezomib plus Pomalidomide and Dexamethasone (Active Comparator)
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Bortezomib

INTERVENTIONS:
Drug: Belantamab mafodotin — Humanized anti-B-cell maturation antigen (BCMA) antibody/drug conjugate will be administered.
  Arms: Arm A: Belantamab mafodotin plus Pomalidomide and Dexamethasone
Drug: Pomalidomide — Immunomodulatory drug (IMiD) will be administered.
Drug: Dexamethasone — Synthetic glucocorticoid with anti-tumor activity will be administered.
Drug: Bortezomib — Proteasome Inhibitor will be administered.
  Arms: Arm B: Bortezomib plus Pomalidomide and Dexamethasone

SUMMARY:
This study will evaluate the efficacy and safety of belantamab mafodotin in combination with pomalidomide and dexamethasone (Arm A) compared with that of combination of pomalidomide, bortezomib and dexamethasone (Arm B) in participants with relapsed/refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent.
* Male or female, 18 years or older.
* Have a confirmed diagnosis of multiple myeloma (MM) as defined by the International Myeloma Working Group (IMWG) criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Have been previously treated with at least 1 prior line of MM therapy including a lenalidomide-containing regimen and must have documented disease progression during or after their most recent therapy. (Participants treated with lenalidomide ≥10 mg daily for at least 2 consecutive cycles are eligible).
* Must have at least 1 aspect of measurable disease defined as one of the following;

  1. Urine M-protein excretion greater than or equal to (≥)200 milligrams (mg) per 24-hour, or
  2. Serum M-protein concentration ≥0.5 grams/deciliters (g/dL) (≥5.0 g/liter [L]), or
  3. Serum free light chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum free light chain ratio (less than [<]0.26 or greater than [>]1.65) only if participant has no measurable urine or serum M spike.
* Have undergone autologous stem cell transplant (ASCT) or are considered transplant ineligible. Participants with a history of ASCT are eligible for study participation provided the following eligibility criteria are met: a. ASCT was >100 days prior to the first dose of study medication. b. No active bacterial, viral, or fungal infection(s) present
* All prior treatment-related toxicities (defined by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI-CTCAE] version 5.0) must be less than or equal to (≤)Grade 1 at the time of enrolment, except for alopecia.
* Adequate organ system functions as mentioned in the protocol.
* Male and female participants agree to abide by protocol-defined contraceptive requirements.

Exclusion Criteria:

* Active plasma cell leukemia, symptomatic amyloidosis or active polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, and skin changes (POEMS) syndrome at the time of screening.
* Prior allogeneic SCT.
* Systemic anti-myeloma therapy (including chemotherapy and systemic steroids) within 14 days or five half-lives (whichever is shorter) preceding the first dose of study drug; prior treatment with a monoclonal antibody drug within 30 days of receiving the first dose of study drugs.
* Plasmapheresis within 7 days prior to the first dose of study drug.
* Received prior treatment with or intolerant to pomalidomide.
* Received prior Beta cell maturation antigen (BCMA) targeted therapy.
* Intolerant to bortezomib or refractory to bortezomib (for example; participant experienced progressive disease during treatment, or within 60 days of completing treatment, with a bortezomib-containing regimen of 1.3 mg/meter square [m^2] twice weekly).
* Evidence of cardiovascular risk including any of the following;

  1. Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram abnormalities including second degree (Mobitz type II) or third degree atrioventricular (AV) block.
  2. Recent history within (3 months of screening) of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting .
  3. Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  4. Uncontrolled hypertension.
* Any major surgery within the last 4 weeks.
* Previous or concurrent invasive malignancy other than multiple myeloma, except:

  1. The disease must be considered medically stable for at least 2 years; or
  2. The participant must not be receiving active therapy, other than hormonal therapy for this disease.
* Known immediate or delayed hypersensitivity reaction or idiosyncratic reaction to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment.
* Evidence of active mucosal or internal bleeding.
* Cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice.
* Active infection requiring treatment.
* Known or active human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C will be excluded unless the protocol-defined criteria are met.
* Presence of active renal conditions (such as infection, severe renal impairment requiring dialysis or any other condition that could affect participant's safety).
* Ongoing Grade 2 peripheral neuropathy with pain within 14 days prior to randomization or ≥Grade 3 peripheral neuropathy.
* Active or history of venous and arterial thromboembolism within the past 3 months.
* Contraindications to or unwilling to undergo protocol-required anti-thrombotic prophylaxis.
* Current corneal disease except for mild punctate keratopathy.
* Any serious and/or unstable pre-existing medical, psychiatric disorder or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures.
* Pregnant or lactating female.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2029-10-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (5):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Nashville, Tennessee
- Australia (11):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Darlinghurst, New South Wales
  - GSK Investigational Site, Gosford NSW, New South Wales
  - GSK Investigational Site, Port Macquarie, New South Wales
  - GSK Investigational Site, Benowa, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Heidelberg, Victoria
  - GSK Investigational Site, Malvern, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Brazil (4):
  - GSK Investigational Site, Curitiba
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, São Paulo
- China (8):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Jiangsu
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Shenyang
  - GSK Investigational Site, Tianjin
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- France (3):
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Vanduvre-lEs-Nancy
- Germany (3):
  - GSK Investigational Site, Mainz
  - GSK Investigational Site, Tübingen
  - GSK Investigational Site, Würzburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Thessaloniki
- Israel (6):
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Tel Aviv
- Italy (4):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Roma
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukushima
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Yamagata
- New Zealand (6):
  - GSK Investigational Site, Auckland
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Grafton
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Takapuna Auckland
  - GSK Investigational Site, Tauranga
- Poland (5):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Wroclaw
- Russia (5):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Sochi
- South Korea (4):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Inchon
  - GSK Investigational Site, Seoul
- Spain (12):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Gijón
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, MOstoles Madrid
  - GSK Investigational Site, Murcia
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, PamplonaNavarra
  - GSK Investigational Site, Pozuelo de AlarcOn Madr
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- Turkey (Türkiye) (5):
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Izmir
  - GSK Investigational Site, Kocaeli
  - GSK Investigational Site, Mersin
  - GSK Investigational Site, Samsun
- United Kingdom (5):
  - GSK Investigational Site, London
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Stoke-on-Trent
  - GSK Investigational Site, Sutton

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

REFERENCES:
- [Derived] Dimopoulos MA, Beksac M, Pour L, Delimpasi S, Vorobyev V, Quach H, Spicka I, Radocha J, Robak P, Kim K, Cavo M, Suzuki K, Wilkes J, McNamara S, Phillips-Jones A, Morris K, Pompilus F, Purser M, Sule N, Kremer B, Loubert A, Bunod L, M'Hari M, Zhou XL, Fulci G, Mateos MV, Trudel S; DREAMM-8 investigators. Patient-reported outcomes with belantamab mafodotin, pomalidomide, and dexamethasone versus bortezomib, pomalidomide, and dexamethasone in patients with relapsed or refractory multiple myeloma (DREAMM-8): a phase 3, open-label, randomised controlled trial. Lancet Haematol. 2025 Nov;12(11):e876-e886. doi: 10.1016/S2352-3026(25)00256-X. PMID 41193117
- [Derived] Hanafin P, Ho YL, Papathanasiou T, Fulci G, Sule N, Kremer BE, Ferron-Brady G. Belantamab Mafodotin with Pomalidomide and Dexamethasone in Relapsed/Refractory Multiple Myeloma: A Comprehensive Exposure-Response Analysis of the DREAMM-8 Study. Target Oncol. 2025 Sep;20(5):833-845. doi: 10.1007/s11523-025-01174-0. Epub 2025 Sep 16. PMID 40958065
- [Derived] Mateos MV, Trudel S, Quach H, Robak P, Beksac M, Pour L, Hus M, Kim K, Zherebtsova V, Delimpasi S, Jelinek T, Ward C, Ho PJ, Vorobyev V, Pitombeira de Lacerda M, Aparecida-Martinez G, Spicka I, Radocha J, Cavo M, Cerchione C, Fu C, Suzuki K, Rogers R, Phillips-Jones A, Wang Z, Baig H, Wilkes J, Zhou XL, Lewis E, Eccersley L, Sule N, Paka P, Opalinska JB, Mukhopadhyay P, Hungria V, Dimopoulos MA. Modification of belantamab mafodotin dosing to balance efficacy and tolerability in the DREAMM-7 and DREAMM-8 trials. Blood Adv. 2025 Nov 25;9(22):5708-5719. doi: 10.1182/bloodadvances.2025016949. PMID 40763276
- [Derived] Dimopoulos MA, Beksac M, Pour L, Delimpasi S, Vorobyev V, Quach H, Spicka I, Radocha J, Robak P, Kim K, Cavo M, Suzuki K, Morris K, Pompilus F, Phillips-Jones A, Zhou XL, Fulci G, Sule N, Kremer BE, Opalinska J, Mateos MV, Trudel S; DREAMM-8 Investigators. Belantamab Mafodotin, Pomalidomide, and Dexamethasone in Multiple Myeloma. N Engl J Med. 2024 Aug 1;391(5):408-421. doi: 10.1056/NEJMoa2403407. Epub 2024 Jun 2. PMID 38828951

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Groups:
- Belantamab Mafodotin+Pomalidomide+Dexamethasone: Participants with Relapsed/Refractory Multiple Myeloma (RRMM) received intravenous (IV) infusion of 2.5 milligram (mg)/kilogram (kg) belantamab mafodotin on Day 1 of Cycle 1 and 1.9 mg/kg on Day 1 of Cycle 2 onwards in each 28-day cycle, in combination with oral 4 mg per day Pomalidomide capsule on Days 1 to 21 of each 28-day cycle; and oral 40 mg per day Dexamethasone tablet on Days 1, 8, 15, and 22 of each 28-day cycle until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of another anti-myeloma therapy or end of study, whichever occurs first.
- Pomalidomide+Bortezomib+Dexamethasone: Participants with RRMM received oral 4 mg per day Pomalidomide capsule on Days 1 to 14 of each 21-day cycle, in combination with subcutaneous (SC) injection of 1.3 mg/meter^2(m^2) Bortezomib on Days 1, 4, 8, 11, of each 21-day cycle for Cycles 1 through 8, and on Days 1, 8, of each 21-day cycle for Cycles 9+, and oral 20 mg Dexamethasone tablet on Days 1, 2, 4, 5, 8, 9, 11, 12, of each 21-day cycle for Cycles 1 through 8 and then on Days 1, 2, 8, 9, every 3 Weeks (Q3W) from Cycles 9 onwards until disease progression, death, unacceptable toxicity, withdrawal of consent, initiation of another anti-myeloma therapy or end of study, whichever occurs first.
Period: Overall Study
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Pomalidomide+Bortezomib+Dexamethasone
Started (Intent-to-Treat (ITT) Population included of all randomized participants whether or not randomized treatment was administered.) | 155 | 147
Safety Population (All randomized participants who received at least 1 dose of study intervention (any component).) | 150 | 145
Completed (Note: Participants who died following randomization whilst on study, were considered to have completed the study.) | 48 (Note: Participants who died following randomization whilst on study, including 1 participant who died prior to dosing.) | 54 (Note: Participants who died following randomization whilst on study, including 1 participant who died prior to dosing.)
Not Completed | 107 | 93
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 11 | 8
Not completed — Ongoing | 94 | 84

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Pomalidomide+Bortezomib+Dexamethasone | Total
Number analyzed (Participants) | 155 | 147 | 302
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 65.5 (8.56) | 66.7 (10.03) | 66.1 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 65 | 121
  Male | 99 | 82 | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (Asian, native Hawaiian OR other pacific islander, and mixed race where 0<n<11) are combined into 'Others' category to maintain participant confidentiality and privacy as the study is evaluating a rare disease.
  Participants
    White | 133 | 127 | 260
    Others | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as time from randomization until earliest date of disease progression (PD), determined by Independent Review Committee (IRC), according to the International Myeloma Working Group (IMWG) Response Criteria, or death due to any cause. PD is defined as increase of >=25% from lowest value in >=1 of following (serum M-protein [absolute increase >=0.5 grams per deciliter {g/dL}]; serum M-protein increase >=1g/dL [when lowest M-protein >=5g/dL]; urine M-protein [absolute increase >=200 milligrams per 24 hours {mg/24h}]; participants without measurable serum & urine M-protein levels, difference between involved & uninvolved serum free light chains (sFLC) levels [absolute increase >10mg/dL]; appearance of new lesion,>=50% increase from nadir in Sum of the products of the maximal perpendicular diameters of measured lesions (SPD) of >1 lesion, or >=50% increase in longest diameter of previous lesion >1 centimeter (cm) in short axis.
Time Frame: Up to approximately 174 weeks
Population: Intent-to-Treat (ITT) Population included all randomized participants whether or not randomized treatment was administered.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Pomalidomide+Bortezomib+Dexamethasone
Number analyzed (Participants) | 155 | 147
Months | NA [20.6 to NA] — NA indicates median and upper limit of 95% CI which were not estimable due to low number of participants with events. | 12.7 [9.1 to 18.5]
Statistical Analysis 1: Comparison: Belantamab Mafodotin+Pomalidomide+Dexamethasone vs Pomalidomide+Bortezomib+Dexamethasone; Test type: Superiority; p < 0.001, Log Rank — P-Value presented to 3 decimal places from one-sided stratified Log-Rank test adjusting for the number of lines of prior therapy (1 vs. 2/3 vs. >=4) and prior bortezomib (yes or no) according to IVRS strata; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.37 to 0.73] — Hazard ratio was estimated using a Cox Proportional Hazards model stratified by the number of lines of prior therapy (1 vs. 2/3 vs. >=4) and prior bortezomib (yes or no) according to IVRS strata with a covariate of treatment

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) defined as the interval of time from randomization to the date of death due to any cause.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

3. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DoR) defined as the time from first documented evidence of PR or better until progressive disease (PD) or death due to any cause. Response will be based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate defined as the percentage of participants who achieve MRD negative status (as assessed by next-generation sequencing at 10^5 threshold) at least once during the time of confirmed CR or better response based on IRC-assessment per IMWG.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

5. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR will be defined as the percentage of participants with a confirmed partial response or better (i.e., PR, VGPR, CR, and sCR) based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

6. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete Response Rate (CRR), defined as the percentage of participants with a confirmed complete response (CR) or better (i.e., CR and stringent complete response (sCR)) based on IRC assessment per IMWG criteria.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

7. Secondary Outcome: Percentage of Participants With a Confirmed Very Good Partial Response (VGPR) or Better
Description: VGPR is defined as the percentage of participants with a confirmed VGPR or better (i.e., VGPR, CR, and sCR) based on IRC-assessment per IMWG criteria.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

8. Secondary Outcome: Time to Best Response (TTBR)
Description: TTBR defined as the interval of time between the date of randomization and the earliest date of achieving best response among participants with a confirmed PR or better based on IRC-assessment per IMWG.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

9. Secondary Outcome: Time to Response (TTR)
Description: TTR defined as the time between the date of randomization and the first documented evidence of response (PR or better) among participants who achieve a response (i.e., confirmed PR or better) based on IRC-assessment per IMWG.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

10. Secondary Outcome: Time to Progression (TTP)
Description: TTP defined as the time from randomization until the earliest date of PD based on IRC-assessment per IMWG criteria, or death due to PD.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

11. Secondary Outcome: Progression-Free Survival 2 (PFS2)
Description: PFS2 defined as time from randomization to disease progression (investigator-assessed response) after initiation of new anti-myeloma therapy or death from any cause, whichever is earlier. If disease progression after new antimyeloma therapy cannot be measured, a PFS event is defined as the date of discontinuation of new anti-myeloma therapy, or death from any cause, whichever is earlier.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

13. Secondary Outcome: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples will be collected for the analysis of hematology parameters.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

14. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples will be collected for the analysis of clinical chemistry parameters.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

15. Secondary Outcome: Number of Participants With Abnormal Ocular Findings on Ophthalmic Examination
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

16. Secondary Outcome: Plasma Concentrations of Belantamab Mafodotin (ADC) at Indicated Time Points
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

17. Secondary Outcome: Plasma Concentrations of Monomethyl Auristatin-F With a Cysteine Linker (Cys-mcMMAF) at Indicated Time Points
Description: Blood samples will be collected for PK analysis of belantamab mafodotin.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

18. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) From Time 0 to the Time of the Last Quantifiable Concentration (C(Tlast)) [AUC (0-last)] for Pomalidomide
Description: Blood samples will be collected for PK analysis of Pomalidomide in combination with belantamab mafodotin and dexamethasone.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

19. Secondary Outcome: Area Under Plasma Concentration-time Curve (AUC) From Time 0 to End of the Dosing Interval [AUC (0-tau)] for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

20. Secondary Outcome: Maximum Concentration (Cmax) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

21. Secondary Outcome: Time of Cmax (Tmax) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

22. Secondary Outcome: Trough Concentration Prior to the Next Dose for Each Cycle (Ctrough) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

23. Secondary Outcome: Last Time Point Where the Concentration is Above the Limit of Quantification (Tlast) for Pomalidomide
Description: as for outcome 18
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

24. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

25. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples will be to be further tested in screening assay, and positive samples will be further characterized for antibody titers.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

26. Secondary Outcome: Number of Participants With Maximum Post-baseline Change From Baseline in Individual Items of Patient-Reported Outcome Version of the Common Term Criteria for Adverse Events (PRO-CTCAE)
Description: The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in participants on cancer clinical trials. The PRO-CTCAE includes an item library of 124 items representing 78 symptomatic toxicities drawn from the CTCAE.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

27. Secondary Outcome: Change From Baseline in Health Related Quality of Life (HRQoL) as Measured by EuropeanOrganization for Research and Treatment of Cancer Quality of Life Questionnaire 30-item Core Module (EORTC QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These includes five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores are averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represents better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represents significant symptomatology. Baseline is defined as latest pre-dose assessment (Day 1) with a non-missing value, including unscheduled visits. Change from Baseline is calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

28. Secondary Outcome: Change From Baseline in Quality of Life Questionnaire 20-item Multiple Myeloma Module (QLQMY20)
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems. A high score for Future Perspective and Body Image represents a high/healthy level of functioning.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

29. Secondary Outcome: Change From Baseline in HRQoL as Measured by EORTC IL52
Description: The EORTC Quality of Life Questionnaire 20-item Multiple Myeloma module (QLQMY20) is a supplement to the QLQ-C30 instrument used in participants with multiple myeloma. For the EORTC IL52, disease symptoms domain of the QLQ-MY20 will be used for bone aches or pain, back pain, hip pain, arm or shoulder pain, chest pain, and pain increasing with activity. The individual component scores in the disease symptom domain are averaged and transformed linearly to a score ranging from 0 to100. A high score for disease symptoms represents a high level of symptomatology or problems. A high score for Future Perspective and Body Image represents a high/healthy level of functioning.
Time Frame: Up to approximately 473 weeks
Reporting Status: Not Posted, anticipated posting 2030-10

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to approximately 174 weeks. The results presented are until the primary completion date. Additional results will be provided within a year of study completion.
Description: Safety population included all randomized participants who receive at least 1 dose of study intervention (any component). Data for All-Cause Mortality was collected for the ITT Population (all randomized participants whether or not randomized treatment was administered). Serious and Other (Not Including Serious) Adverse Events were collected for the Safety Population (all randomized participants who received at least 1 dose of study intervention [any component]).
Arm/Group | Belantamab Mafodotin+Pomalidomide+Dexamethasone | Pomalidomide+Bortezomib+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 48/155 | 54/147
Serious Adverse Events (participants affected / at risk) | 95/150 | 65/145
Other Adverse Events (participants affected / at risk) | 148/150 | 130/145
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin+Pomalidomide+Dexamethasone (N=150) | Pomalidomide+Bortezomib+Dexamethasone (N=145)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (6) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 9 (13) | 4 (4)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (6)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3)
Cardiac failure (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (2)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 3 (3)
Device related thrombosis (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 10 (10) | 4 (5)
COVID-19 pneumonia (Infections and infestations) | 17 (18) | 6 (7)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 2 (2)
Klebsiella infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 1 (1)
Parvovirus B19 infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 (5) | 0 (0)
Pneumonia (Infections and infestations) | 27 (33) | 11 (11)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (6) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Varicella (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Visceral leishmaniasis (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Craniofacial fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (5) | 4 (4)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belantamab Mafodotin+Pomalidomide+Dexamethasone (N=150) | Pomalidomide+Bortezomib+Dexamethasone (N=145)
Anaemia (Blood and lymphatic system disorders) | 35 (52) | 37 (63)
Neutropenia (Blood and lymphatic system disorders) | 69 (206) | 48 (191)
Thrombocytopenia (Blood and lymphatic system disorders) | 54 (113) | 40 (99)
Cataract (Eye disorders) | 40 (56) | 14 (16)
Corneal epithelial microcysts (Eye disorders) | 34 (51) | 0 (0)
Corneal opacity (Eye disorders) | 13 (23) | 0 (0)
Dry eye (Eye disorders) | 91 (232) | 14 (17)
Eye irritation (Eye disorders) | 75 (198) | 13 (16)
Eye pain (Eye disorders) | 49 (100) | 7 (7)
Foreign body sensation in eyes (Eye disorders) | 91 (257) | 9 (12)
Keratitis (Eye disorders) | 8 (9) | 1 (1)
Keratopathy (Eye disorders) | 11 (14) | 0 (0)
Lacrimation increased (Eye disorders) | 9 (11) | 4 (4)
Photophobia (Eye disorders) | 66 (168) | 6 (6)
Punctate keratitis (Eye disorders) | 34 (63) | 1 (1)
Vision blurred (Eye disorders) | 119 (426) | 22 (24)
Visual acuity reduced (Eye disorders) | 34 (62) | 8 (11)
Visual impairment (Eye disorders) | 23 (54) | 2 (2)
Constipation (Gastrointestinal disorders) | 22 (35) | 33 (42)
Diarrhoea (Gastrointestinal disorders) | 34 (56) | 32 (50)
Nausea (Gastrointestinal disorders) | 18 (28) | 15 (16)
Asthenia (General disorders) | 15 (26) | 20 (29)
Fatigue (General disorders) | 40 (45) | 32 (39)
Oedema peripheral (General disorders) | 16 (21) | 23 (26)
Pyrexia (General disorders) | 28 (41) | 9 (11)
Hypogammaglobulinaemia (Immune system disorders) | 8 (10) | 6 (7)
Bronchitis (Infections and infestations) | 11 (14) | 6 (10)
COVID-19 (Infections and infestations) | 48 (57) | 27 (30)
Infection (Infections and infestations) | 3 (7) | 8 (10)
Nasopharyngitis (Infections and infestations) | 9 (15) | 7 (13)
Pneumonia (Infections and infestations) | 13 (15) | 9 (10)
Upper respiratory tract infection (Infections and infestations) | 39 (64) | 25 (46)
Urinary tract infection (Infections and infestations) | 20 (36) | 13 (16)
Alanine aminotransferase increased (Investigations) | 23 (34) | 13 (23)
Aspartate aminotransferase increased (Investigations) | 15 (20) | 11 (15)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 6 (6)
Blood creatinine increased (Investigations) | 9 (10) | 5 (14)
Gamma-glutamyltransferase increased (Investigations) | 10 (15) | 3 (3)
Neutrophil count decreased (Investigations) | 30 (116) | 19 (100)
Platelet count decreased (Investigations) | 30 (55) | 21 (40)
Decreased appetite (Metabolism and nutrition disorders) | 9 (10) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 11 (12) | 10 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 11 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (20) | 21 (27)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (8)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 (15) | 8 (10)
Dizziness (Nervous system disorders) | 9 (9) | 17 (20)
Headache (Nervous system disorders) | 9 (10) | 8 (13)
Neuropathy peripheral (Nervous system disorders) | 11 (16) | 34 (44)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 15 (22)
Tremor (Nervous system disorders) | 9 (10) | 5 (6)
Insomnia (Psychiatric disorders) | 20 (23) | 18 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 11 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (9) | 10 (14)
Rash (Skin and subcutaneous tissue disorders) | 11 (13) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT04484623/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-02): https://cdn.clinicaltrials.gov/large-docs/23/NCT04484623/SAP_001.pdf